CLINICAL TRIAL: NCT02299960
Title: Pilot Study: Analysis of Endothelial Function Through Circulating Endothelial Cells and Puls-amplitude-tonometry and of Non-invasive Measurement of Cardiac Output on Exertion in Patients With Heart Failure, Pulmonary Hypertension, Arterial Hypertension and Diabetic Nephropathy
Brief Title: Measurement of Endothelial Function and Cardiac Output: New Methods
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Bayer (Industry); Health Twist GmbH (Unknown)
Responsible Party: Principal Investigator, Sebastian Beckmann, Doctoral candidate, Charite University, Berlin, Germany
Other Study IDs: ENDO-CEC
Record Dates: First submitted 2014-11-20; First posted 2014-11-24 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-06

CONDITIONS: Heart Failure; Hypertension, Pulmonary; Hypertension; Diabetic Nephropathies
Keywords: EndoPAT; NICOM; circulating endothelial cells
MeSH Terms: conditions — Heart Failure; Hypertension, Pulmonary; Hypertension; Diabetic Nephropathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples, 51,4ml per Patient

GROUPS / COHORTS (4):
- HFpEF: patients with heart failure with preserved ejection fraction
  Interventions: Device: Endo-PAT; Device: NICOM
- HFrEF: patients with heart failure with reduced ejection fraction
  Interventions: Device: Endo-PAT
- AH: patients with hypertension
  Interventions: Device: Endo-PAT; Device: NICOM
- Nephropathy: patients with diabetic nephropathy
  Interventions: Device: Endo-PAT

INTERVENTIONS:
Device: Endo-PAT — Analysis of endothelial function through pulse-amplitude-tonometry
Device: NICOM — Non-invasive measurement of cardiac output
  Groups: AH; HFpEF

SUMMARY:
The main purpose of this study is to analyse test-retest-reliability of functional quantification of endothelial dysfunction through puls-amplitude-tonometry in patients with heart failure with preserved/reduced ejection fraction, pulmonary hypertension, arterial hypertension and diabetic nephropathy. In the same group, test-retest-reliability of circulating endothelial cells as well as test-retest reliability of non invasive cardiac output Monitoring will be observed and analysed.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable for the last 4 weeks (not for HFrEF: 7 days)
* Signed consent form

HFpEF:

* Baseline-Echocardiography:
* hospitalization <= 12 months with diagnosis heart failure and E/E' > 8 or E' < 8 cm/s or
* BNP >= 100pg/ml or NT-proBNP >= 300pg/ml in the last 6 months or
* LAVI > 28 ml/m² and E/E' > 8 or E' < 8cm/s or PAPsys > 40mmHg and E/E' > 8 or E' < 8 cm/s
* Possibility to take part in cardiac stress test
* Heart failure NYHA I-III
* Sinus rhythm
* Max. O2-uptake on exertion < 20ml/kgBW/min

HFrEF

* HFrEF due to ischemic or non-ischemic reasons
* NYHA I-III
* Individually optimized and stable pharmacological therapy (including beta-blocker, ACE-Inhibitor, AT1-antagonist, aldosterone-antagonist)
* EF <=45%, Simpson Biplan PH
* NICE-Classification 2013 I/II
* PAH >= 25 mmHg
* Precapillary PAH: Wedge-pressure <= 15 mmHg, CO normal or low
* Postcapillary PAH: Wedge-pressure >= 15 mmHg, CO normal or low

Diabetic nephropathy:

* Diabetes mellitus Type 2 with oral or Insulin therapy and one or more of the following:
* Diabetic nephropathy has been diagnosed before (anamnesis)
* Macroalbuminuria: Urine Albumine/Creatinine-ratio > 300mg/g Creatinine (>34mg/mmol) in 2 out of 3 tests of Urine in the morning and GFR <90ml/min/1.73m² (CKD-EPI)
* Microalbuminuria: 30-300mg/g Creatinine (>=3.4 mg/mmol but <34mg/mmol) tested as above and GFR < 90 ml/min/1.73m² and diabetic retinopathy

AH:

* Hypertension diagnosed at least 6 months except structural heart disease: EF > 55% and no sign of HFpEF
* No symptoms of coronary heart disease
* Possibility to take part in cardiac stress test
* Stable pharmacologic therapy of Hypertension for at least 4 weeks
* Systolic blood pressure <140 mmHG during Screening

Exclusion Criteria:

* Patient incapable of contracting
* Angina pectoris > CCS II
* Coronary Intervention in the last 4 weeks or scheduled Intervention/Bypass
* Myocardial infarction in the last 3 months
* Stroke in the last 3 months
* Valvular heart disease > II°
* Cardiomyopathy due to Infiltrate/hypertrophic obstruction (e.g. HOCM, Amyloidosis)
* Congenital complex heart disease
* Active myocarditis
* Significant lung disease
* Significant Cardiac dysrhythmia
* Scheduled changes in medication during time of study
* (Scheduled) heart transplant
* Cardiac resynchronisation therapy over the last three months
* ICD/Pacemaker-implant in the last 4 weeks
* Uncontrolled Hyper/Hypotension (>180mmHg, <95mmHg)
* Patient taking part in Rehabilitation program
* Diagnosed Malignant disease or disease with life expectancy < 1 year
* Anemia with Hb<10mg/dl
* Untreated significant thyroid disease

HFpEF, Hypertension and PH:

* Patient incapable of cardiac stress test (e.g. because of orthopedic Problems)
* Significant changes in cardiovascular Status over the two weeks of study
* Instable cardiopulmonary Status over the last four weeks

HFrEF:

* I.v. Treatment with inotropic drug or diuretic in the last 7 days before Screening
* Myocardial infarction in the last 4 weeks

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from the conditions stated above
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2014-08; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Test-retest-reliability EndoPAT | 2 weeks

SECONDARY OUTCOMES:
Test-retest-reliability circulating endothelial cells | 2 weeks
Test-retest-reliability NICOM | 2 weeks
Correlation: Cardiac Output on exertion and cardiopulmonary exercise test and 6 Minute Walking test | 2 weeks
Correlation: circulating endothelial cells and EndoPAT and endothelial function | 2 weeks
  will include the molecular diagnostic of circulating endothelial cells
Variability of biomarkers of myocardiac remodelling and of cardiorenal syndrome | 2 weeks
Correlation cardiac Output on exertion and echocardiography in HFpEF | 2 weeks
Clinical feasibility of circulating endothelial cells and EndoPAT | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Dirk Duengen, PD Dr. med., Study Chair — Charite Universitaetsmedizin Berlin
Locations (1):
- Charite Universitaetsmedizin, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Weisrock F, Fritschka M, Beckmann S, Litmeier S, Wagner J, Tahirovic E, Radenovic S, Zelenak C, Hashemi D, Busjahn A, Krahn T, Pieske B, Dinh W, Dungen HD. Reliability of peripheral arterial tonometry in patients with heart failure, diabetic nephropathy and arterial hypertension. Vasc Med. 2017 Aug;22(4):292-300. doi: 10.1177/1358863X17706752. Epub 2017 May 30. PMID 28555533